CLINICAL TRIAL: NCT04658576
Title: Pre-operative Ultrasonographic Evaluation of Caval Aorta Diameter Index as a New Predictor for Hypotension After Induction of General Anaesthesia: A Prospective Observational Cohort Study.
Brief Title: Pre-operative Ultrasonographic Evaluation of Caval Aorta Diameter Index as a Predictor for Post-induction Hypotension
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shymaa Fathy, Lecturer of anesthesia and SICU, Cairo University
Other Study IDs: MD-245-2020
Record Dates: First submitted 2020-12-02; First posted 2020-12-08 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Hypotension on Induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Comparison between ultrasound measurement of IVCD-AOd index in prediction of post induction hypo tension

DETAILED DESCRIPTION:
This study aims to evaluate the ability of preoperative ultrasound measurements IVC to aorta diameter index to predict post-induction hypotension in comparison with ultrasound measurements of the IVC collapsibility index.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients (>18years)

  * ASA I-II

Exclusion Criteria:

* • ASA physical status > II

  * Dyspnea
  * Systolic blood pressure ≥ 180 mmHg
  * Systolic blood pressure < 90 mmHg
  * Agitation (RASS > 1)
  * IVC non visualized
  * Epidural catheter in use
  * Patients with increased intraabdominal pressure (intrabdominal mass compressing IVC).
  * Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: • Patients scheduled for elective orthopedic surgeries under general anaesthesia
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-10-23 (Actual); Study Completion 2022-10-23 (Actual)

PRIMARY OUTCOMES:
• Comparison of the accuracy Area under receiver operating characteristic curves (AUROC) of IVCD:AoD index and IVCCI in prediction of post-induction hypotension | 15 minutes
  Measurement of pre-operative IVC-AOrta diameter index and IVC collapsibility index

CONTACTS AND LOCATIONS:
Overall Officials: Shymaa Fathy, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No